CLINICAL TRIAL: NCT06452979
Title: Mucosal Inflammation in Children With OSA - Potential Biomarkers of OSA Complications
Brief Title: Mucosal Inflammation in Children With OSA
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kate Ching Ching Chan, Associate Professor, Chinese University of Hong Kong
Other Study IDs: MOSA
Record Dates: First submitted 2023-11-01; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Biological samples including nasal epithelial lining fluid and blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Children aged 6-11 years old with habitual snoring (≥3 nights per week) and PSG confirmed OSA (OAHI of ≥1/hour)
- Controls: Non-OSA age, sex and BMI-matched control with PSG confirmed absence of OSA (OAHI < 1 event/h)

SUMMARY:
Objectives: Variability of clinical phenotypes in childhood obstructive sleep apnoea (OSA) has prompted research for biomarkers to identify patients at risk of developing OSA-related complications. Upper airway inflammation is documented in children with OSA. Whether it is related to end-organ morbidities and systemic inflammation is under-explored. The primary objectives of our study are 1)To evaluate inflammatory biomarkers with the use of nasal epithelial lining fluid (NELF) collected by nasal strips as a representation of upper airway inflammation in children with OSA compared to non-OSA controls; 2) To evaluate the associations between NELF biomarkers with ambulatory blood pressure (ABP) outcomes in children with OSA.

Hypothesis to be tested: Inflammatory biomarkers in NELF in children with OSA are altered when compared with non-OSA controls and correlated with ABP outcomes.

Design and subjects: A prospective case-control study. Non-obese Chinese children aged 6-11 years old with habitual snoring (≥3 nights per week) and polysomnography (PSG) confirmed OSA (OAHI of ≥1/hour) will be recruited as cases. Non-OSA children with OAHI < 1 event/h will be recruited as controls. All subjects will undergo evaluation including questionnaires, anthropometric measurements, PSG, 24-hour ABP measurement, blood and NELF sampling.

Primary outcome measure: Profile of inflammatory biomarkers in the NELF. Analysis: Correlations between NELF inflammatory biomarkers with polysomnographic and ABP measurements will be evaluated by regression analysis.

Expected results: This study will provide novel and important information regarding upper airway inflammatory biomarkers in children with OSA and their relationship with blood pressure outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-11 years old

Exclusion Criteria:

* Previous upper airway surgery, genetic or syndromal disease, congenital or acquired neuromuscular disease, suspected or confirmed congenital or acquired immunodeficiency, obesity (BMI z-score ≥1.645), known metabolic syndrome, craniofacial abnormalities, structural or congenital heart disease, use of medications or therapy that could affect immunity such as systemic corticosteroids, chemotherapy, radiation therapy, intravenous immunoglobulins.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Chinese children aged 6-11 years old with symptoms suggestive of obstructive sleep apnoea and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Inflammatory profile in the nasal fluid | 3 years
  Profile of inflammatory biomarkers in the nasal epithelial lining fluid: cytokines profiles

SECONDARY OUTCOMES:
Inflammatory profile in the peripheral blood | 3 years
  Systemic inflammatory biomarkers collected from peripheral blood: cytokines profiles

CONTACTS AND LOCATIONS:
Overall Officials: Kate Ching Ching Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong